CLINICAL TRIAL: NCT01026740
Title: An Exploratory Study to Evaluate the Penetration of Ceftobiprole Into Soft Tissue Determined by In Vivo Microdialysis in Healthy Volunteers
Brief Title: Evaluation of Penetration of Ceftobiprole Into Soft Tissue Determined by Microdialysis in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Basilea Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CR011416; CSI-1002 (Other: Basilea)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Staphylococcal Skin Infections; Streptococcal Infections
Keywords: Staphylococcal Skin Infections; Streptococcal Infections
MeSH Terms: conditions — Staphylococcal Skin Infections; Streptococcal Infections | interventions — ceftobiprole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 001 (Experimental): Ceftobiprole 500 mg, single infusion over 2 hours
  Interventions: Drug: Ceftobiprole

INTERVENTIONS:
Drug: Ceftobiprole — single intravenous (i.v.) infusion, 500 mg ceftobiprole administered over 2 hours.

SUMMARY:
The primary objective of this study is to measure the penetration of ceftobiprole into subcutaneous (s.c.) adipose tissue and skeletal muscle and to determine the concentration over time of ceftobiprole in these tissues and in plasma after administration of a single intravenous (i.v.) infusion (directly into the vein) of ceftobiprole 500 mg administered over 2 hours. The secondary objective was to further assess the safety and tolerability of ceftobiprole after a single i.v. infusion.

DETAILED DESCRIPTION:
This is a single-center, open-label (all patients involved know the identity of the drug), single-arm, nonrandomized study of ceftobiprole in healthy men and women. The study is conducted in 2 parts: a pilot study and a main study. Each study (i.e. the pilot study and the main study) consists of 3 phases: a pretreatment phase that includes up to a 21-day screening period, an open-label treatment phase (1 day in the pilot study and 2 days in the main study), and a posttreatment phase that included the end of study evaluations and follow-up study visit or telephone contact planned for 1 to 2 weeks after discharge from the study unit. Serial blood and dialysis samples will be collected at specified time points from predose through 24 hours after the start of the infusion for estimation of ceftobiprole and ceftobiprole medocaril concentrations. Additional samples will be collected for measurement of protein binding. The study will include the following evaluations of safety and tolerability: adverse events, clinical laboratory tests (including hematology, serum chemistry, and urinalysis), electrocardiogram (ECG), vital signs, physical examination, serology, pregnancy tests, urine drug screen, and alcohol breath test. In the pilot study, Ceftobiprole will be locally administered via a microdialysis probe at a concentration of approximately 30 µg/mL for 60 minutes. In the main Study, each volunteer will receive ceftobiprole locally via the microdialysis probe. After the washout period determined by the pilot study, each volunteer will receive a single 2-hour i.v. infusion of ceftobiprole.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI between 18 to 29 kg/m2
* Nonsmoker
* Normal renal function

Exclusion Criteria:

* History of gastric or duodenal ulcer
* History of allergies or hypersensitivity (including penicillin, cephalosporins, or other ß-lactams or quinolones)
* Hypersensitivity or intolerance to heparin
* History of drug or alcohol abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2007-06; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
To measure the penetration of ceftobiprole into subcutaneous (s.c.) adipose tissue and skeletal muscle and to determine the concentration-versus-time profiles of ceftobiprole in these tissues and in plasma. | Day 1 pre- and post-dose during the pilot study and on Days 1 and 2 during the main study

SECONDARY OUTCOMES:
To assess the safety and tolerability of ceftobiprole after a single intravenous (iv) infusion. | Approximately 5 weeks during the pilot study including screening, treatment, and posttreatment follow up and for approximately 5 weeks during the main study including screening, treatment, and posttreatment follow up

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An Exploratory Study to Evaluate the Penetration of Ceftobiprole Into Soft Tissue Determined by In Vivo Microdialysis in Healthy Volunteers — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=732&filename=CR011416_REF1.pdf
- See also: An Exploratory Study to Evaluate the Penetration of Ceftobiprole Into Soft Tissue Determined by In Vivo Microdialysis in Healthy Volunteers — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=732&filename=CR011416_CSR.pdf